CLINICAL TRIAL: NCT04938258
Title: Feasibility and Potential Effectiveness of a Case Management Intervention for Alcohol Use-Related Problems in Frequent Users of an Emergency Department: a Pilot Study
Acronym: MALUA_Freq_P
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual rate to achieve expected sample size.
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Hugo López-Pelayo, MD, PhD, IDIBAPS Grup de Recerca en Addiccions Clinic Emeritus Researcher, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2019/0717 ER-01; HCB/2019/0717 ER-01 (Other: Hospital Clínic de Barcelona Ethics Committee)
Record Dates: First submitted 2021-06-04; First posted 2021-06-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Drinking; Alcohol-Related Disorders
MeSH Terms: conditions — Alcohol Drinking; Alcohol-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive Case Management Intervention (Experimental): Participants will receive an intensive Case Management (CM) intervention conducted by a multidisciplinary team during 2 months. They will attend weekly or biweekly appointments with the CM team, the interviews will last approximately 30 minutes and will be conducted based on Motivational Interviewing techniques in order to explore values and needs and to enhance motivation to reduce alcohol use and self-efficacy.
  Receiving the CM intervention doesn't exclude treatment as usual.
  Interventions: Behavioral: Intensive Case Management

INTERVENTIONS:
Behavioral: Intensive Case Management — Participants will receive an intensive Case Management (CM) intervention conducted by a multidisciplinary team (Psychiatry, Social Work, Nursing) during 2 months. The intervention will encompass attending weekly or biweekly appointments with the CM team, the interviews will last approximately 30 minutes. This CM intervention will include referral to Hospital Clínic de Barcelona Addiction Outpatient Clinic and a personalised assessment of the medical, psychiatric and social situation of each individual by the CM team. An individualised care plan will be established and periodically reviewed by the multidisciplinary team in response to a better understanding of patient needs or to a change in patient health condition. The intervention will offer motivational interviewing psychotherapy to enhance motivation to reduce or to quit alcohol use, in crisis intervention, coordination of care, patient education and self-management support, and assistance to navigate in the healthcare system.

SUMMARY:
Alcohol use and its consequences represent an important public health problem. As well as alcohol dependence, hazardous drinking also contributes to a high burden in terms of morbidity and mortality. To improve these patients' prognosis and decrease associated social and health care costs, it is necessary to increase early detection, intervention and treatment for these problems. Alcohol consumption is associated with a decrease in primary care services utilization, thus Emergency Departments (EDs) are a primary gateway to healthcare services in this group.

Depending on the investigative method and the mixture of the target population, an estimated 0.6-40% of all ED visits are due to alcohol-related problems. Given this, EDs offer a unique window of opportunity to address alcohol problems.

The threshold most commonly used to define frequent use of EDs is more than 4 visits per year. Frequent users comprise 0.3% to 10% of all ED patients and account for 3.5% to 28% of ED visits in developed countries. Addictive and other psychiatric disorders, and also social vulnerability are more common in frequent ED users than in non-frequent users. Although case management interventions seem promising to reduce ED attendance among frequent users, currently there is mixed evidence on the effects of such interventions on ED use.

Considering all this, a broader understanding of interventions to reduce frequent visits is needed, specially focusing on local frequent ED populations and identified highly vulnerable subgroups, such as hazardous drinkers.

The investigators aim to evaluate the feasibility and potential effectiveness of a Case Management programme for ED Frequent Users presenting risky alcohol use in the ED of a tertiary hospital.

DETAILED DESCRIPTION:
Methods:

Unicentric, national, open, non-controlled pre-post pilot study to evaluate the feasibility and potential effectiveness of a Case Management programme for ED Frequent Users presenting risky alcohol use in the ED of a tertiary hospital in Barcelona. All patients between 18 and 65 years old that frequently attended Hospital Clínic of Barcelona emergency department during the previous year that reattend the ED during the recruitment period will be eligible to follow-up. Those of them presenting risky alcohol use according to AUDIT-C score that consent to participate will receive a case management intervention as well as treatment as usual. Main outcomes will be change in the number of visits to the ED and change in proportion of risky drinkers measured by AUDIT-C at 12 months follow-up.

Case management (CM) can be defined as a collaborative process of assessment, planning, facilitation, and advocacy for options and services to meet an individual's health needs through communication and available resources to promote quality cost-effective outcomes. Case managers identify appropriate providers and services for individual patients while simultaneously ensuring that available resources are being used in a timely and cost-effective manner. It is a model of continuous, integrated medical and psychosocial care, which is markedly different from the episodic and often fragmented care that occurs in the ED setting. Close partnerships with healthcare providers and community services resources are key factors of CM interventions, that should target patients with the greatest needs.

ELIGIBILITY:
Inclusion Criteria:

* 5 or more attendances during the previous 12 months at the Emergency Department of Hospital Clínic de Barcelona
* an AUDIT-C score higher than 5 points for men and 4 for women
* Patients who accept to participate in the study and give informed consent
* Exists valid contact information to reach patient in the future.

Exclusion Criteria:

* There is psychopathology that prevents study comprehension and/or future participation (i.e. cognitive impairment, acutely psychotic, acutely confused, intoxicated...)
* Patients who present medical conditions that predict that will not be able to participate in follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in number of Emergency Department Visits | At 12 months after enrollment
  Change compared to previous year
Change from baseline in the proportion of risky drinkers measured by AUDIT-C (Alcohol Use Disorders Identification Test-Consumption) | At 12 months after enrollment
  Participants will be assessed with AUDIT-C (a tool to assess alcohol consumption). Main outcome 2 is the proportion of patients who score more than 5 in men and more than 4 in women in this scale.
  Minimum value: 0. Maximum value: 12. Higher scores indicate more severity of alcohol use.
Change from baseline in the severity of alcohol use according to AUDIT (Alcohol Use Disorders Identification Test) score (as a continuous variable) | At 12 months after enrollment
  Minimum value: 0. Maximum value: 40. Higher scores indicate more severity of alcohol use.

SECONDARY OUTCOMES:
Change from baseline in quality of life according to EQ-5D-5L questionnaire descriptive system (5-digit number that describes the patient's health state) | At 12 months after enrollment
  The EQ-5D-5L (5-level EQ-5D version (EQ-5D-5L) by the EuroQol Group) is a generic test to assess quality of life related to health. It includes 5 dimensions of quality of life (mobility, self-care, daily activities, pain, anxiety/depression) as a description of the patient's health state. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change from baseline in quality of life according to EQ-5D-5L questionnaire visual analogue scale (EQ VAS): patient's self-rated health from 0 to 100 | At 12 months after enrollment
  The EQ-5D-5L (5-level EQ-5D version (EQ-5D-5L) by the EuroQol Group) is a generic test to assess quality of life related to health. It includes the EQ VAS, which records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled from score 100 ('The best health you can imagine') to 0 ('The worst health you can imagine'). The VAS can be used as a quantitative measure of health outcome.
Change from baseline in psychiatric symptoms severity through Brief Psychiatric Rating Scale (BPRS) | At 12 months after enrollment
  BPRS is a clinician rating scale that provides an assessment of common psychopathology symptoms. Minimum value: 18. Maximum value: 126. Higher scores indicate more severity of psychiatric symptoms.
Change from previous year in number of hospital admissions | At 12 months after enrollment
  Need of inpatient care

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gual, PhD, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams S, Brown A, Patton R, Crawford MJ, Touquet R. The half-life of the 'teachable moment' for alcohol misusing patients in the emergency department. Drug Alcohol Depend. 2005 Feb 14;77(2):205-8. doi: 10.1016/j.drugalcdep.2004.07.011. PMID 15664722
- [Background] Vu F, Daeppen JB, Hugli O, Iglesias K, Stucki S, Paroz S, Canepa Allen M, Bodenmann P. Screening of mental health and substance users in frequent users of a general Swiss emergency department. BMC Emerg Med. 2015 Oct 9;15:27. doi: 10.1186/s12873-015-0053-2. PMID 26452550
- [Background] Simioni N, Rolland B, Cottencin O. Interventions for Increasing Alcohol Treatment Utilization Among Patients with Alcohol Use Disorders from Emergency Departments: A Systematic Review. J Subst Abuse Treat. 2015 Nov;58:6-15. doi: 10.1016/j.jsat.2015.06.003. Epub 2015 Jun 23. PMID 26206477
- [Background] Klein LR, Driver BE, Miner JR, Martel ML, Cole JB. Emergency department length of stay for ethanol intoxication encounters. Am J Emerg Med. 2018 Jul;36(7):1209-1214. doi: 10.1016/j.ajem.2017.12.017. Epub 2017 Dec 8. PMID 29305022
- [Background] Klein LR, Martel ML, Driver BE, Reing M, Cole JB. Emergency Department Frequent Users for Acute Alcohol Intoxication. West J Emerg Med. 2018 Mar;19(2):398-402. doi: 10.5811/westjem.2017.10.35052. Epub 2018 Feb 26. PMID 29560072
- [Background] Urbanoski K, Cheng J, Rehm J, Kurdyak P. Frequent use of emergency departments for mental and substance use disorders. Emerg Med J. 2018 Apr;35(4):220-225. doi: 10.1136/emermed-2015-205554. Epub 2018 Jan 8. PMID 29311114
- [Background] Verelst S, Moonen PJ, Desruelles D, Gillet JB. Emergency department visits due to alcohol intoxication: characteristics of patients and impact on the emergency room. Alcohol Alcohol. 2012 Jul-Aug;47(4):433-8. doi: 10.1093/alcalc/ags035. Epub 2012 Apr 5. PMID 22493048
- [Background] Anderson P, Berridge V, Conrod P, Dudley R, Hellman M, Lachenmeier D, Lingford-Hughes A, Miller D, Rehm J, Room R, Schmidt L, Sullivan R, Ysa T, Gual A. Reframing the science and policy of nicotine, illegal drugs and alcohol - conclusions of the ALICE RAP Project. F1000Res. 2017 Mar 17;6:289. doi: 10.12688/f1000research.10860.1. eCollection 2017. PMID 28435669
- [Background] Bruguera P, Barrio P, Oliveras C, Braddick F, Gavotti C, Bruguera C, Lopez-Pelayo H, Miquel L, Segura L, Colom J, Ortega L, Vieta E, Gual A. Effectiveness of a Specialized Brief Intervention for At-risk Drinkers in an Emergency Department: Short-term Results of a Randomized Controlled Trial. Acad Emerg Med. 2018 May;25(5):517-525. doi: 10.1111/acem.13384. Epub 2018 Apr 2. PMID 29418049
- [Background] Bruguera P, Barrio P, Manthey J, Oliveras C, Lopez-Pelayo H, Nuno L, Miquel L, Lopez-Lazcano A, Blithikioti C, Caballeria E, Matrai S, Rehm J, Vieta E, Gual A. Mid and long-term effects of a SBIRT program for at-risk drinkers attending to an emergency department. Follow-up results from a randomized controlled trial. Eur J Emerg Med. 2021 Oct 1;28(5):373-379. doi: 10.1097/MEJ.0000000000000810. PMID 33709997
- [Background] Locker TE, Baston S, Mason SM, Nicholl J. Defining frequent use of an urban emergency department. Emerg Med J. 2007 Jun;24(6):398-401. doi: 10.1136/emj.2006.043844. PMID 17513534
- [Background] Bieler G, Paroz S, Faouzi M, Trueb L, Vaucher P, Althaus F, Daeppen JB, Bodenmann P. Social and medical vulnerability factors of emergency department frequent users in a universal health insurance system. Acad Emerg Med. 2012 Jan;19(1):63-8. doi: 10.1111/j.1553-2712.2011.01246.x. Epub 2012 Jan 5. PMID 22221292
- [Background] LaCalle E, Rabin E. Frequent users of emergency departments: the myths, the data, and the policy implications. Ann Emerg Med. 2010 Jul;56(1):42-8. doi: 10.1016/j.annemergmed.2010.01.032. Epub 2010 Mar 26. PMID 20346540
- [Background] Meng X, Muggli T, Baetz M, D'Arcy C. Disordered lives: Life circumstances and clinical characteristics of very frequent users of emergency departments for primary mental health complaints. Psychiatry Res. 2017 Jun;252:9-15. doi: 10.1016/j.psychres.2017.02.044. Epub 2017 Feb 21. PMID 28237761
- [Background] Moschetti K, Iglesias K, Baggio S, Velonaki V, Hugli O, Burnand B, Daeppen JB, Wasserfallen JB, Bodenmann P. Health care costs of case management for frequent users of the emergency department: Hospital and insurance perspectives. PLoS One. 2018 Sep 24;13(9):e0199691. doi: 10.1371/journal.pone.0199691. eCollection 2018. PMID 30248102
- [Background] Moe J, Kirkland S, Ospina MB, Campbell S, Long R, Davidson A, Duke P, Tamura T, Trahan L, Rowe BH. Mortality, admission rates and outpatient use among frequent users of emergency departments: a systematic review. Emerg Med J. 2016 Mar;33(3):230-6. doi: 10.1136/emermed-2014-204496. Epub 2015 May 7. PMID 25953837
- [Background] Giannouchos TV, Kum HC, Foster MJ, Ohsfeldt RL. Characteristics and predictors of adult frequent emergency department users in the United States: A systematic literature review. J Eval Clin Pract. 2019 Jun;25(3):420-433. doi: 10.1111/jep.13137. Epub 2019 May 2. PMID 31044484
- [Background] Shumway M, Boccellari A, O'Brien K, Okin RL. Cost-effectiveness of clinical case management for ED frequent users: results of a randomized trial. Am J Emerg Med. 2008 Feb;26(2):155-64. doi: 10.1016/j.ajem.2007.04.021. PMID 18272094
- [Background] Althaus F, Paroz S, Hugli O, Ghali WA, Daeppen JB, Peytremann-Bridevaux I, Bodenmann P. Effectiveness of interventions targeting frequent users of emergency departments: a systematic review. Ann Emerg Med. 2011 Jul;58(1):41-52.e42. doi: 10.1016/j.annemergmed.2011.03.007. PMID 21689565
- [Background] Kumar GS, Klein R. Effectiveness of case management strategies in reducing emergency department visits in frequent user patient populations: a systematic review. J Emerg Med. 2013 Mar;44(3):717-29. doi: 10.1016/j.jemermed.2012.08.035. Epub 2012 Nov 29. PMID 23200765
- [Background] Moe J, Kirkland SW, Rawe E, Ospina MB, Vandermeer B, Campbell S, Rowe BH. Effectiveness of Interventions to Decrease Emergency Department Visits by Adult Frequent Users: A Systematic Review. Acad Emerg Med. 2017 Jan;24(1):40-52. doi: 10.1111/acem.13060. PMID 27473387
- [Background] Hudon C, Chouinard MC, Lambert M, Diadiou F, Bouliane D, Beaudin J. Key factors of case management interventions for frequent users of healthcare services: a thematic analysis review. BMJ Open. 2017 Oct 22;7(10):e017762. doi: 10.1136/bmjopen-2017-017762. PMID 29061623
- [Background] Kahan D, Poremski D, Wise-Harris D, Pauly D, Leszcz M, Wasylenki D, Stergiopoulos V. Perceived Case Management Needs and Service Preferences of Frequent Emergency Department Users: Lessons Learned in a Large Urban Centre. PLoS One. 2016 Dec 21;11(12):e0168782. doi: 10.1371/journal.pone.0168782. eCollection 2016. PMID 28002491
- [Background] Parkman T, Neale J, Day E, Drummond C. How Do People Who Frequently Attend Emergency Departments for Alcohol-Related Reasons Use, View, and Experience Specialist Addiction Services? Subst Use Misuse. 2017 Sep 19;52(11):1460-1468. doi: 10.1080/10826084.2017.1285314. Epub 2017 May 3. PMID 28467154